CLINICAL TRIAL: NCT05434130
Title: Modulating Exercise Dosage to Improve Concussion Recovery: a Randomized Clinical Trial
Brief Title: Modulating Exercise Dosage to Improve Concussion Recovery
Acronym: MEDIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Boston Children's Hospital (Other); Spaulding Rehabilitation Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-4932; R01HD108133 (NIH)
Record Dates: First submitted 2022-05-26; First posted 2022-06-27 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Concussion, Brain; Treatment; Aerobic Exercise; Inflammation; Depression, Anxiety
Keywords: intervention; mild traumatic brain injury
MeSH Terms: conditions — Brain Concussion; Inflammation; Depression; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study will use a block stratified RCT design. Our stratum factors are the biological variable of sex and recruitment location
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study PI, Co-Is, and the biostatistician will not know group assignments until after the primary analyses are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Dose Exercise (Experimental): The investigators will provide exercise dose recommendations for initial visit until symptom resolution, and revise upon symptom resolution (to use for the subsequent 8 weeks). These include intensity (target HR) and volume (frequency/duration). Intensity is calculated as 90% of the HR at the end of the exercise test. The volume recommendation is 150 mins/week (~30 min/day; 5 days/week). The mode of exercise is another consideration. This will be left to participant preference, so that the investigators do not exclude potential participants due to lack of access to specific exercise equipment.
  Interventions: Behavioral: High Dose Exercise
- Standard-of-care (No Intervention): Participants are instructed to perform activity in line with physician recommendations. This consists of a general recommendation (no specific HR/volume) or symptom limited physical activity.

INTERVENTIONS:
Behavioral: High Dose Exercise — The investigators will initially test and randomize adolescents ages 13-18 years old ≤14 days post-concussion to high dose aerobic exercise (>150 min/week, individualized intensity level) or standard-of-care (symptom limited, self-guided physical activity), and re-test upon symptom resolution and 8-weeks post symptom resolution
  Arms: High Dose Exercise

SUMMARY:
Aerobic exercise has emerged as an effective treatment to reduce sport-related concussion symptom severity, yet existing work lacks rigor regarding the precise exercise volume and intensity required to elicit therapeutic effects, how exercise can alter concussion-related pathophysiology, and whether exercise can prevent the development of secondary sequelae. Our objective is to examine if a high dose exercise program (higher volume than currently prescribed at an individualized, safe intensity level) initiated within 14 days of concussion results in faster symptom resolution, altered physiological function, or reduced secondary sequalae. Findings from this research will lead to more rigorous and precise rehabilitation guidelines and improved understanding about how exercise affects neurophysiological function among adolescents with concussion.

DETAILED DESCRIPTION:
Concussions are defined as a mild form of traumatic brain injury that result in acute neurological dysfunction. Recent work suggests post-concussion aerobic exercise at an intensity level below symptom exacerbation is safe. Yet, clinical benefits from existing randomized controlled trials indicate substantial room for improvement. Also, there is currently an incomplete understanding of the neurophysiology underlying changes in response to exercise treatment. Identifying the precise exercise dose (volume/intensity) required to elicit a therapeutic response following concussion will lead to enhanced and more precise post-concussion rehabilitation strategies. Published and pilot data by the investigators indicate light post-concussion exercise was associated with faster symptom resolution time and less severe symptoms, yet this relied on self-reported data and observational designs. Furthermore, the investigators have identified that the optimal exercise volume to differentiate those with/without concussion symptoms after one month was >160 minutes/week, which is higher than standard exercise volumes prescribed (>100 minutes/week), and in line with existing recommendations for cardiovascular health (>150 minutes/week). Beyond this, given the positive effects of regular moderate exercise to reduce inflammation (e.g., interleukin 6) and restore cerebrovascular regulation, these physiological functions represent viable and feasible rehabilitation targets. Thus, using a prospective randomized clinical trial design, the investigators aim to identify if high dose exercise >(150 minutes/week at an individualized intensity level), relative to standard-of-care, results in: faster/slower symptom resolution, altered physiological function, or reduced secondary sequalae. Our multidisciplinary investigative team has expertise investigating concussion, exercise physiology, fluid biomarkers, cerebrovascular physiology, and psychosocial outcomes. Thus, the investigators will enroll, initially test, and randomize adolescents ages 13-18 years old ≤14 days post-concussion to high dose aerobic exercise or standard-of-care (symptom limited, self-guided physical activity), and reassess upon symptom resolution and 8-weeks post symptom resolution. The investigators will obtain cerebrovascular function and serum biomarker data at each visit, and quantify exercise, symptoms, and secondary sequalae continuously. First, The investigators aim to examine how the dose (intensity, duration, and frequency) of an aerobic exercise program initiated within 10 days of concussion affects time to symptom resolution, relative to standard-of-care, among adolescents. Second, the investigators aim to assess the mechanistic relationship between aerobic exercise, biomarkers of neuroinflammation, and cerebrovascular function. Third, the investigators aim to elucidate how high dose exercise after concussion affects persistent secondary sequalae development (anxiety, depression, kinesiophobia, peer relationships, academic concerns). By challenging the currently accepted, exercise recommendations for sport-related concussion, the investigators will break new ground toward improving rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years of age
* Post-Concussion Symptom Scale (PCSS) score >10 to ensure participants are not recovered by enrollment
* Concussion diagnosis by a sports medicine physician

Exclusion Criteria:

* Pre-existing neurological disorders
* Exercise contraindications
* Concussion <6 months before enrollment (excluding the current injury)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Time from injury to symptom resolution | From time of injury until defined symptom resolution observed, about 30 days
  The PCSS is a standard form that records the presence and severity of 22 concussion symptoms at the time of testing. Participants rate their concussion symptoms from 0-6 where 0 equates to "no symptoms," and 6 to "severe symptoms."
Serum biomarker concentration: GFAP change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  Concentrations of GFAP will be simultaneously assayed along with other biomarkers using multi-plex digital array technology, which allows for single molecule immunoarrays while minimizing the amount of sample required
Anxiety and depression severity change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  Participants will report anxiety using the Hospital Anxiety and Depression Scale (HADS).The HADS addresses questions related to depression and anxiety symptoms. Responses range from 0 to 3, where 3=experiencing symptoms a great deal of the time, on 14 questions. Seven items are specific to depression symptoms, and 7 to anxiety symptoms. For each sub-scale (HADS-anxiety and HADS-depression) scores range from 0 (no symptoms) to 21 (maximum symptom severity).

SECONDARY OUTCOMES:
Serum biomarker concentration: IL-6 change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  Concentrations of IL-6 will be simultaneously assayed along with other biomarkers using multi-plex digital array technology, which allows for single molecule immunoarrays while minimizing the amount of sample required
Serum biomarker concentration: TNF-alpha change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  Concentrations of TNF-alpha will be simultaneously assayed along with other biomarkers using multi-plex digital array technology, which allows for single molecule immunoarrays while minimizing the amount of sample required
Serum biomarker concentration: IL1-RA change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  Concentrations of IL1-RA will be simultaneously assayed along with other biomarkers using multi-plex digital array technology, which allows for single molecule immunoarrays while minimizing the amount of sample required
Serum biomarker concentration: VEGF change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  Serum biomarkers will be obtained via venipuncture at the initial visit, after symptom resolution, and 8 weeks after symptom resolution.
Serum biomarker concentration: MMP-9 change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  Concentrations of MMP-9 will be simultaneously assayed along with other biomarkers using multi-plex digital array technology, which allows for single molecule immunoarrays while minimizing the amount of sample required
Cerebral autoregulation | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  The investigators will examine the ability to buffer against pressure changes during exercise. Autoregulation will be assessed by deriving the relationship between arterial pressure and cerebral blood flow fluctuations elicited using low resistance breathing.
Cerebral vasoreactivity change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  The investigators will examine the ability to increase blood flow in response to increases in blood CO2. This is assessed by measuring the progressive increase in cerebral blood flow in response to progressive increases in inspired CO2.
Kinesiophobia severity change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  The Tampa Scale of Kinesiophobia (TSK) is a 17-item self-report, 4-point Likert scale questionnaire designed to assess fear of pain with movement (kinesiophobia). The questionnaire was originally designed to measure fear of pain during movement among patients with low back pain, and is reliable.
Peer relationship attitudes change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  Using the Patient Reported Outcomes Measurement Information System (PROMIS), The investigators will obtain data regarding participant attitudes toward peer relationships (friends and other acquaintances).
Academic concerns change | Baseline, Visit 2 (scheduled after symptoms resolve, about 35 days post-baseline)
  The Concussion Learning Assessment and School Survey (CLASS) aims to assess concern for the effect of concussion on school learning, new or exacerbated post-concussion academic problems, and perceived impact on academic performance.

CONTACTS AND LOCATIONS:
Overall Officials: David R Howell, PhD, Principal Investigator — University of Colorado Denver | Anschutz
Locations (3):
- United States (3):
  - University of Colorado Denver, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Spaulding Rehabilitation Hospital, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No